CLINICAL TRIAL: NCT06079385
Title: The Effect of Acupuncture Treatment on Sleep Quality in Post-Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstPRMTRH3
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Complementary
Keywords: acupuncture; sleep medicine; stroke
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): The patients who received acupuncture treatment in addition to a standard rehabilitation program
  Interventions: Other: Acupuncture treatment
- Control group (No Intervention): The patients who received the standard rehabilitation program.

INTERVENTIONS:
Other: Acupuncture treatment — Acupuncture treatment with needles
  Arms: Acupuncture group

SUMMARY:
The aim of this study is to investigate the effectiveness and reliability of acupuncture treatment in patients experiencing impaired sleep quality after a stroke. Additionally, the goal is to reduce the need for multiple medications and/or high-dose drug usage in the treatment of these complications in patients

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of acupuncture therapy on sleep quality in patients experiencing insomnia in the early post-stroke period. In this prospective, randomized controlled, single-blind study, 70 ischemic stroke patients undergoing inpatient rehabilitation were included. Participants were randomly divided into two groups: the acupuncture group receiving acupuncture therapy and standard rehabilitation program. The control group receiving only the standard rehabilitation program. The acupuncture group received acupuncture treatment twice a week for 4 weeks. Sleep quality was evaluated using the Pittsburgh Sleep Quality Index (PSQI). The PSQI scores were assessed three times at baseline, at the 4th week, and at the 8th week. The results of the study indicated that the acupuncture group demonstrated a significant improvement in sleep quality compared to the control group. Significant differences were observed between the baseline PSQI scores and the PSQI scores at the 4th week in both the acupuncture and control groups (p: 0.000 and p: 0.008). The change between baseline and 8th-week PSQI scores was also significant (p: 0.000 and p: 0.000). However, in the acupuncture group, the decrease in PSQI scores was significantly greater compared to the control group. The addition of acupuncture therapy to standard treatment resulted in a significant improvement in sleep quality. Additionally, the baseline PSQI scores were found to be correlated with the severity of depression.This study suggests that acupuncture therapy can be an effective intervention for improving sleep quality in patients with early post-stroke insomnia.

ELIGIBILITY:
Inclusion Criteria:

* being between 18-80 years of age,
* having a minimum of 2 and a maximum of 6 months elapsed since the ischemic stroke, -volunteering to participate in the study,
* having a mini-mental test score above 17.

Exclusion Criteria:

* history of insomnia or depression before stroke,
* psychiatric medication use,
* psychiatric illness, aphasia, sleep apnea syndrome,
* decompensated cardiac, renal, or hepatic insufficiency, pregnancy,
* presence of infection in the areas where acupuncture would be applied.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 0 day, 4th week and 8th week
  The index helps to evaluate sleep quality of patient. The scores range from 0 to 21 and the authors suggest that a score >5 be considered as a significant sleep disturbance.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | 0 day, 4th week and 8th week
  The scale is used to evaluate symptoms related to depression. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale
Hamilton Anxiety Rating Scale | 0 day, 4th week and 8th week
  The scale is used to evaluate symptoms related to anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Barthel Index | 0 day
  it helps to evaluate the patient's functional status. scores of 0-20 indicate "total" dependency scores of 21-60 indicate "severe" dependency scores of 61-90 indicate "moderate" dependency scores of 91-99 indicate "slight" dependency
Mini-Mental State Examination | 0 day
  the test is used to evaluate patient's cognitive status. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age

CONTACTS AND LOCATIONS:
Overall Officials: Nur Kesiktas, MD, Prof, Study Chair — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao H, Pan X, Li H, Liu J. Acupuncture for treatment of insomnia: a systematic review of randomized controlled trials. J Altern Complement Med. 2009 Nov;15(11):1171-86. doi: 10.1089/acm.2009.0041. PMID 19922248
- [Background] Xiang J, Li H, Xiong J, Hua F, Huang S, Jiang Y, Zhou X, Liao K, Xu L. Acupuncture for post-stroke insomnia: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Jul 24;99(30):e21381. doi: 10.1097/MD.0000000000021381. PMID 32791749
- [Background] Niu S, Liu X, Wu Q, Ma J, Wu S, Zeng L, Shi Y. Sleep Quality and Cognitive Function after Stroke: The Mediating Roles of Depression and Anxiety Symptoms. Int J Environ Res Public Health. 2023 Jan 29;20(3):2410. doi: 10.3390/ijerph20032410. PMID 36767777
- [Result] Lee SH, Lim SM. Acupuncture for insomnia after stroke: a systematic review and meta-analysis. BMC Complement Altern Med. 2016 Jul 19;16:228. doi: 10.1186/s12906-016-1220-z. PMID 27430619